CLINICAL TRIAL: NCT04969107
Title: Abdominal or Transanal TME in Therapy of Rectal Cancer: A Retrospective Cohort Study
Brief Title: Abdominal or Transanal TME for Rectal Cancer Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Lukas Marti, Dr. med. Lukas Marti, Leitender Arzt Chirurgie, Cantonal Hospital of St. Gallen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMEabdVSta
Record Dates: First submitted 2021-06-11; First posted 2021-07-20 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Survival; Postoperative Morbidity; Mortality; Recurrence
Keywords: TME; Rectal Cancer; transanal; local recurrence
MeSH Terms: conditions — Recurrence; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- transanal TME (taTME) (Active Comparator): patients with rectal cancer receiving transanal TME
  Interventions: Procedure: taTME
- abdominal TME (abTME) (Active Comparator): patients with rectal cancer receiving open, laparoscopic or robotic TME
  Interventions: Procedure: abdTME

INTERVENTIONS:
Procedure: taTME — Resection of rectal cancer with preparation of the mesorectal plane along the TME-plane in a rendezvous procedure of an abdominal and a transanal approach.
  Other Names: transanal total mesorectal excision
  Arms: transanal TME (taTME)
Procedure: abdTME — Resection of rectal cancer with preparation of the mesorectal plane along the TME-plane in an abdominal Approach.
  Other Names: abdominal total mesorectal excision
  Arms: abdominal TME (abTME)

SUMMARY:
This study assessed whether transanal TME in patients with rectal cancer is superior to open, laparoscopic, and robotic TME (abdominal TME (abTME)) regarding oncological outcome, postoperative morbidity and 90-day mortality.

DETAILED DESCRIPTION:
Rectal cancer accounts for 3.8% of all new cancer diagnosis and for 3.4% of all cancer-related deaths in the world in 2020. Regarding treatment of rectal cancer, it is essential to perform surgery along the anatomical and embryological planes. This technique called total mesorectal excision (TME) reduces the local recurrence rate and improves the survival. Since the early 2000, TME has changed from open to laparoscopic approach due to better results in short-term outcome. Nevertheless, oncological benefits are modest. In 2009 the first ever transanal TME (taTME) war performed. This novel technique combines abdominal with transanal dissection. Because the distal part of the rectum is approached from below, a better visualization of the mesorectal plane resulting in higher rate of free CRM and of complete TME specimen grade (Quirke Score) can be accomplished. However, taTME remains a hot topic in the current scientific literature. In Norway and the Netherlands a higher rate of anastomotic leakage as well as a higher rate of local recurrence (9.5%) with multifocal growth pattern were described.

ELIGIBILITY:
Inclusion Criteria:

* all patients receiving elective total mesorectal excision

Exclusion Criteria:

* diagnosis other than rectal cancer
* partial mesorectal excision
* discontinuity resection (no anastomosis)
* incomplete Staging
* metastatic cancer
* lack of follow-up
* decline of a retrospective data Analysis
* age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 60 months
  time from surgery to end of follow-up or death
cancer-specific survival | 60 months
  time from surgery to end of follow-up or death due to rectal cancer
disease-specific survival | 60 months
  time from surgery to end of follow-up or death due to or recurrence of rectal cancer

SECONDARY OUTCOMES:
positive resection margin | 30 days
  tumor extending to the resection margin in pathological examination (R0, R1)
Quirke Score | 30 days
  Quality of mesorectal excision in pathological examination (Good, modest, bad)
circular resection margin (CRM) | 30 days
  size of circular resection margin (mm) in pathological examination
number of lymph nodes | 30 days
  number of lymph nodes in pathological examination
postoperative morbidity | 30 days
  Number of patients with postoperative complications (bleeding, anastomotic leakage, ileus, sacral infect, fistula, other surgical complications). The complications will be classified according the Clavien-Dindo-Classification
postoperative 90-day mortality | 90 days
  Number of patients who die in the first 90 days after surgery
relapse-free survival | 60 months
  local recurrence
recurrence-free survival | 60 months
  local or systemic recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Marti, Dr. med., Study Director — Leitender Arzt, Chirurige KSSG
Locations (1):
- Department of surgery, Cantonal hospital of St. Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No